CLINICAL TRIAL: NCT00612781
Title: Influence of Blue-Light-Filter IOLs on Color Perception and Contrast Acuity. A Randomized, Double-Masked Study With Intraindividual Comparison.
Brief Title: Yellow Versus White Study
Acronym: YeWhi
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Hietzing (Other)
Responsible Party: Matthias Wirtitsch MD, Dept. of Ophthalmology, Hospital Hietzing, Vienna, Austria
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ye-Whi 2006
Record Dates: First submitted 2008-01-29; First posted 2008-02-12 (Estimated); Last update posted 2008-02-12 (Estimated); Status verified 2008-01

CONDITIONS: Cataract
Keywords: intraocular lens; blue-light filtering intraocular lens; contrast acuity; color vision
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Other)
  Interventions: Procedure: cataract surgery (Hoya AF-1 [UY] YA-60BB)
- B (Other)
  Interventions: Procedure: cataract surgery (Hoya AF-1 [UV] VA-60BB lens)

INTERVENTIONS:
Procedure: cataract surgery (Hoya AF-1 [UY] YA-60BB) — implantation of a yellow Hoya AF-1 (UY) YA-60BB intraocular lens
  Other Names: Hoya AF-1 (UY) YA-60BB
  Arms: A
Procedure: cataract surgery (Hoya AF-1 [UV] VA-60BB lens) — implantation of an uncoloured Hoya AF-1 (UV) VA-60BB
  Other Names: Hoya AF-1 (UV) VA-60BB
  Arms: B

SUMMARY:
Blue-light-filtering IOLs are implanted increasingly often in cataract surgery. Several studies examined the effect of blue-light-filters on contrast and colour vision. However, the study outcomes were varying. The present study investigated the effect of a blue-light-filtering IOL on colour perception and contrast acuity using highly sensitive measurement methods.

ELIGIBILITY:
Inclusion Criteria:

* bilateral age-related cataract
* age 55 to 80 years
* expected postoperative visual acuity of at least 1.0

Exclusion Criteria:

* amblyopia
* corneal scars
* diabetes
* arterial hypertonia
* pseudoexfoliation-syndrome
* earlier ocular surgeries or laser treatments
* intraocular tumors
* color abnormalities
* expected postoperative visual acuity lower 1.0

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-12; Primary Completion 2007-02 (Actual); Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
contrast sensitivity | 3 month after surgery
color vision | 3 month after surgery

SECONDARY OUTCOMES:
visual acuity | 3 month after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Matthias G Wirtitsch, MD, Principal Investigator — Dept of Ophthalmology, Hietzing Hospital, Vienna, Austria
Locations (1):
- Department of Ophthalmology, Hietzing Hospital, Vienna, Austria